CLINICAL TRIAL: NCT00164385
Title: Adolescent Impact: A Behavioral Intervention for Adolescents Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3723; U64CCU219448; U64CCU319455; U64CCU319459
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: Adolescent Impact

SUMMARY:
The primary objective of Adolescent Impact is to develop and evaluate a developmentally targeted intervention designed to minimize secondary transmission risk behavior and enhance adherence to care and treatment. The intervention is delivered in 12 sessions (five one-to-one, 7 group) over a 3 month period of time. Intervention is delivered in addition to standard of care treatment at the participant's respective clinic. Participants are randomized to either an intervention or control arm; the control group receives standard of care treatment and control group participants are offered the Adolescent Impact intervention following the completion of the nine-month follow up. It is hypothesized that compared to control group participants, intervention group participants will evidence (1) improved or stable virologic and/or immunologic status, mediated by (a) adherence to prescribed antiretroviral medication and/or (b) adherence to HIV care appointments, and (2) reduction/minimization of secondary transmission risk behaviors to include (a) unprotected sex and/or needle sharing, and (b) sexual and drug use behaviors that increase risk for unprotected sex.

DETAILED DESCRIPTION:
The primary objective of Adolescent Impact is to develop and evaluate a developmentally targeted intervention designed to minimize secondary transmission risk behavior and enhance adherence to care and treatment. The intervention is delivered in 12 sessions (five one-to-one, 7 group) over a 3 month period of time. Intervention is delivered in addition to standard of care treatment at the participant's respective clinic. Participants are randomized to either an intervention or control arm; the control group receives standard of care treatment and control group participants are offered the Adolescent Impact intervention following the completion of the nine-month follow up. It is hypothesized that compared to control group participants, intervention group participants will evidence (1) improved or stable virologic and/or immunologic status, mediated by (a) adherence to prescribed antiretroviral medication and/or (b) adherence to HIV care appointments, and (2) reduction/minimization of secondary transmission risk behaviors to include (a) unprotected sex and/or needle sharing, and (b) sexual and drug use behaviors that increase risk for unprotected sex.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection
2. Followed at one of the participating clinics for HIV care
3. Age 13-21 at enrollment (i.e., must be enrolled prior to 22nd birthday)
4. Aware of HIV status and, for perinatally infected teens, the HIV status of one's biological mother
5. Able to comprehend English well enough to participate in the study
6. Able to understand and sign a written informed consent or assent
7. Parental or legal guardian consent, if under the age of 18 -

Exclusion Criteria:

1. Less than borderline intellectual functioning, as evidenced by clinician assessment or full scale IQ less than 65
2. Acute and severe mental illness (including, but not limited to, psychosis, severe depression, or significant suicidal or homicidal ideation) -

Ages: 13 Years to 21 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Koenig, PhD, Study Chair — Centers for Disease Control and Prevention